CLINICAL TRIAL: NCT00073801
Title: The Neural Immune Mechanisms and Genetic Influences on Chronic Pelvic Pain in Women With Endometriosis
Brief Title: Pelvic Pain in Women With Endometriosis
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040056; 04-N-0056
Record Dates: First submitted 2003-12-08; First posted 2003-12-09 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Endometriosis; Chronic Pelvic Pain
Keywords: Myofascial Dysfunction; Sensitization; Healthy Volunteers; Overlapping Pain Conditions; Hypothalamic-Pituitary-Adrenal Axis; Natural History
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic Pelvic Pain and Endometriosis: Women with chronic pelvic pain and endometriosis found at study surgery
- Chronic Pelvic Pain and No Endometriosis: Women with chronic pelvic pain and NO endometriosis found at study surgery
- Healthy Volunteers: Women without no chronic pelvic pain and no symptoms of endometriosis

SUMMARY:
This study will examine pelvic pain associated with endometriosis and explore better approaches to treatment. In women with endometriosis, uterine tissue grows outside the uterus. Standard treatments - altering hormone levels to prevent endometrial tissue growth or surgically removing endometrial tissue - treat pelvic pain only temporarily. This study will investigate the role of sex hormones, immune chemicals, stress hormones, and genes in pelvic pain and determine how the nerve, muscle, and skeletal systems are involved in this pain.

Women between 18 and 50 years of age who:

1. have endometriosis and chronic pelvic pain, and
2. have chronic pelvic pain without endometriosis, and
3. have neither endometriosis nor chronic pelvic pain and are willing to have a tubal ligation (Healthy Volunteer group),

may be eligible for this study. Candidates are screened with a questionnaire to obtain information about their pain and previous treatments and related medical or social issues. Participants will undergo the following tests and procedures:

1. Medical history and physical examination, including pelvic exam, blood tests, urinalysis, and diaphragm fitting.
2. Questionnaires about pain, quality of life, sexuality, psychological attitudes, spiritual experiences, and history of headache and depression.
3. At-home monitoring for 4 to 6 weeks of pain symptoms, menstruation and spotting, medicines taken, and urine collections to test for "LH" surge. LH is the hormone that causes the ovary to release a mature egg.
4. Pre-laparoscopy evaluation to include:

   * Examination of menstrual blood collected in a diaphragm for 4 hours.
   * Blood sampling to measure adrenal and pituitary hormones. For this test, corticotrophin-releasing hormone (CRH) is injected through an IV needle. Up to five blood samples are drawn, starting before the injection until 45 minutes after it. Blood is also collected at this time for genetic analysis.
   * In-depth pain assessment to identify trigger points in muscles associated with pelvic pain, regions of skin sensitivity, and bone pain. Some women will undergo microdialysis, which uses an acupuncture-type needle to collect chemicals from two different muscles.
   * Blood sampling twice a week for 1 month to measure changes in blood substances during the menstrual cycle.
   * Blood sampling after the LH surge to measure progesterone levels.
   * Cervicovaginal lavage (washing of the cervix with saline and collecting the fluid) to obtain secretions for research.
   * Ultrasound of the ovaries and uterus. This examination uses a probe inserted into the vagina that emits sound waves that are used to form pictures of the internal structures. A small piece of uterine lining is also obtained for examination and research purposes.
   * A visit with the members of the Pain and Palliative care service to evaluate the pain in anticipation of offering other treatments for pain after surgery.
   * Surgery:

CPP + Endo or CPP only: Laparoscopy to look for and remove endometrial tissue. This procedure is done under general anesthetic. A viewing instrument called a laparoscope is passed through an incision in the belly button to look for endometriosis. If it is found, two or more incisions are made in the abdomen for other instruments to remove the tissue. A small piece of uterine lining is also obtained for examination and research purposes.

Healthy Volunteers: Laparoscopy to perform the tubal ligation. A tubal ligation, commonly known as "getting your tubes tied," is a surgical procedure for women to sterilize them. This procedure closes the fallopian tubes, stopping the egg from traveling from the ovary to the uterus and preventing sperm from reaching the fallopian tube to fertilize an egg. In a tubal ligation, fallopian tubes are cut, burned, or blocked with rings, bands or clips. The surgery is effective immediately. Tubal ligations are 99.5% effective as birth control. This procedure is done under general anesthetic. A viewing instrument called a laparoscope is passed through an incision in the belly button to perform a tubal ligation. Two or more incisions are made in the abdomen for other instruments to perform the procedure. During the laparoscopy, we will look for and remove endometrial tissue. A small piece of uterine lining is also obtained for examination and research purposes.

-Follow-up evaluations. Two weeks after surgery, patients return to NIH to discuss the surgical findings and treatment options. Follow-up visits are then scheduled at 1, 3, and 6 months after surgery to complete questionnaires and determine if the treatment is working. Blood samples are drawn at each visit.

DETAILED DESCRIPTION:
Chronic pelvic pain associated with endometriosis is poorly understood. This study is an effort to better understand pelvic pain and identify novel medical approaches for treating it. Endometriosis is a very common disease of women in their reproductive years, in which endometrial tissue grows outside the uterus. In a recent epidemiologic study, we have shown strong associations among endometriosis, fibromyalgia, and autoimmune disorders. Currently, it is believed that endometriosis causes chronic pelvic pain. Yet, some women with endometriosis do not have any pain and others have pain in areas unrelated to endometriosis disease location. The standard approaches to treating endometriosis pain have been to medically alter hormone levels to prevent endometriosis tissue growth or to surgically remove endometriosis lesions. Pelvic pain is only temporarily treated by either approach, which suggests that the current classification of pain, based on disease and treatment with hormones or surgery is not adequate. The feeling of pain involves many complex processes. Generally, women suffer more frequently from chronic, long-term, painful conditions than men. This suggests that women process pain differently because of differences in sex hormone levels and genes expressed in a sexually dimorphic fashion, as well as in central nervous and immune system function differences. We will examine the relations among sex hormones, pain processing, immune system substances and pain related genes. We will also examine changes in levels of hormonal and immune substances in the blood, endometriosis lesions and normal endometrial tissue. Myofascial pain has been noted in women with endometriosis and chronic pelvic pain. We will study how the nerve, muscle and skeletal systems are involved in pelvic pain by performing an in depth pain assessment. Finally, stress plays an important role generating and perpetuating chronic pain. We will examine how the hormones related to the stress response may be altered in pelvic pain.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women between the ages of 18 and 50 years, who have their reproductive organs. Those undergoing tubal ligation must be at least 21 years old.

Excellent health other than a three-month history of pelvic pain and documented endometriosis at laparoscopy. Chronic medications may be acceptable at the discretion of the Principal Investigator (PI). Use of antidepressants, medications for migraines and headaches, allergy medications, and treatment of bowel symptoms such as irritable bowel disease will be allowed.

Do not desire pregnancy for the duration of the study.

Are using abstinence, mechanical (condoms, diaphragms) or sterilization methods of contraception and are willing to continue using them throughout the study.

Willing and able to give informed consent.

Willing and able to comply with study requirements.

BMI < than 32 kg/m^2.

History of regular cyclic menses.

EXCLUSION CRITERIA:

Women with other causes of chronic pelvic pain including infectious, gastrointestinal, psychologic disorders, fibromyalgia and chronic fatigue syndrome.

Significant abnormalities in the physical or laboratory examination including renal and liver function more than twice the normal range.

Hysterectomy or bilateral salpingo-oophorectomy.

Pregnancy.

Lactation.

Use of hormonal contraception, selective estrogen receptor modulators, progestins, estrogens, steroids, or ovulation induction in the last 3 months.

Other medical or surgical treatment for endometriosis in the last 6 months.

Untreated abnormal pap smear or other gynecologic condition.

Manic-depressive illness or untreated major depression.

HIV infection.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We plan to study women of reproductive age with chronic pelvic pain, some of whom have endometriosis and some who do not. Healthy women without chronic pelvic pain and not known to have endometriosis will serve as controls. In the event that endometriosis is found at laparoscopy in the control group, we will include these patients in the study as a separate subset of controls. Controls may choose to complete the study, including laparoscopy with a tubal ligation, complete the study without laparoscopy, or participate in an abbreviated study that includes only screening and chronic stress testing. All women will be protected from pregnancy by non-hormonal contraception such as barrier contraception, abstinence or surgical sterilization for the duration of the study.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2004-04-22 (Actual)

PRIMARY OUTCOMES:
To evaluate the menstrual dynamics of systemic cytokine expression in endometriosis, and to measure the expression of pro-inflammatory cytokines, stem cells, immunologic activity, and neurotransmittors in endometriosis lesions and the endometriu... | Day 1-3 of the menstrual cycle; by twice weekly blood draws between 8 and 9 AM (14 ml/time) over a four-week period; Mid-luteal cervical secretions and endometrium
  menstrual effluent by collecting menses over a four- hour period on day one to three of the menstrual cycle; Menstrual cycle variation in systemic secretion of inflammatory mediators (IL-6) and hormones, estradiol and progesterone;Mid-luteal cervical secretions and endometrium for measurement of pro and anti-inflammatory effectors

SECONDARY OUTCOMES:
To evaluate the relation between chronic pelvic pain and the HPA axis in women | Follicular phase of the menstrual cycle
  CRH stimulation testing. The HPA assessments will include the measurement of morning levels of serum ACTH and cortisol and the serum levels of ACTH and cortisol after CRH stimulation test.
To evaluate whether routine Pain and Palliative Care services of medication adjustment, psychosocial and spiritual counseling, and mind- body techniques offered post- operatively contribute to relief from pain | post-operative over six months
  analysis of records from Pain and Palliative care
To investigate the influence of genetic polymorphisms in pain pathways, pro-inflammatory cytokines, and mediators of sensitization on chronic musculoskeletal pain in women. | preoperative evaluation
  linkage association and with haplotype mapping genomic on DNA that was freshly isolated and stored at 70 degrees C
to quantitatively and qualitatively characterize the musculoskeletal components of chronic pelvic pain associated with endometriosis by a standardized neuromusculo-skeletal evaluation. | Follicular phase of the menstrual Cycle
  Identification of myofascial trigger points in muscles associated with pelvic pain and use pressure algometry to measure pressure pain threshold (the minimal pressure that causes pain; Identification of regions of cutaneous allodynia using Semmes-Weinstein monofilaments across abdominal and pelvic dermatomes. Identification of regions of cutaneous hyperalgesia with a Wartenberg pinwheel across abdominal and pelvic dermatomes. Identification of regions of periosteal tenderness using pressure algometry over bony prominences.

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Al-Harthi L, Spear GT, Hashemi FB, Landay A, Sha BE, Roebuck KA. A human immunodeficiency virus (HIV)-inducing factor from the female genital tract activates HIV-1 gene expression through the kappaB enhancer. J Infect Dis. 1998 Nov;178(5):1343-51. doi: 10.1086/314444. PMID 9780254
- [Background] Al-Harthi L, Wright DJ, Anderson D, Cohen M, Matity Ahu D, Cohn J, Cu-Unvin S, Burns D, Reichelderfer P, Lewis S, Beckner S, Kovacs A, Landay A. The impact of the ovulatory cycle on cytokine production: evaluation of systemic, cervicovaginal, and salivary compartments. J Interferon Cytokine Res. 2000 Aug;20(8):719-24. doi: 10.1089/10799900050116426. PMID 10954915
- [Background] Berkley KJ. Sex differences in pain. Behav Brain Sci. 1997 Sep;20(3):371-80; discussion 435-513. doi: 10.1017/s0140525x97221485. PMID 10097000
- [Derived] Stratton P, Khachikyan I, Sinaii N, Ortiz R, Shah J. Association of chronic pelvic pain and endometriosis with signs of sensitization and myofascial pain. Obstet Gynecol. 2015 Mar;125(3):719-728. doi: 10.1097/AOG.0000000000000663. PMID 25730237
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-N-0056.html